CLINICAL TRIAL: NCT00006026
Title: Open Label Phase II Study on RFS 2000 (9-Nitro-Camptothecin, 9-NC) Administered as a "5 Days On-2 Days Off" Oral Treatment in Advanced/Metastatic Urothelial Tract Tumors
Brief Title: Nitrocamptothecin in Treating Patients With Metastatic Cancer of the Urinary Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16996U; EORTC-16996U
Record Dates: First submitted 2000-07-05; First posted 2004-03-16 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: recurrent bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder; squamous cell carcinoma of the bladder; adenocarcinoma of the bladder; recurrent urethral cancer; anterior urethral cancer; posterior urethral cancer; urethral cancer associated with invasive bladder cancer; metastatic transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — rubitecan

INTERVENTIONS:
Drug: rubitecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of nitrocamptothecin in treating patients who have metastatic cancer of the urinary tract.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response to nitrocamptothecin in patients with metastatic urothelial tract tumors. II. Determine the response rate in these patients when treated with this regimen. III. Determine the duration of objective response in these patients when treated with this regimen. IV. Characterize the toxicities of this treatment in this patient population.

OUTLINE: This is a multicenter study. Patients receive oral nitrocamptothecin daily on days 1-5. Treatment continues weekly every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 weeks until disease progression.

PROJECTED ACCRUAL: A total of 14-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic or unresectable primary carcinoma of the urinary tract including bladder, ureter, and renal pelvis Transitional cell carcinoma OR Mixed cell carcinoma OR Squamous cell carcinoma OR Adenocarcinoma Measurable disease At least 20 mm by conventional techniques OR At least 10 mm by spiral CT scan No symptomatic brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) Alkaline phosphatase and transaminases no greater than 2.5 times ULN (no greater than 5 times ULN in case of hepatic metastases) Renal: Creatinine no greater than 1.7 mg/dL Cardiovascular: Normal cardiac function No ischemic disease in past 6 months Other: Not pregnant or nursing Fertile patients must use effective contraception No other prior malignancies except cone biopsied carcinoma of the cervix or adequately treated basal or squamous cell skin carcinoma No concurrent unstable systemic disease or active uncontrolled infection No psychological, familial, sociological, or geographical condition that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Must have received 1 prior chemotherapy regimen for advanced or metastatic disease At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: At least 14 days since prior major surgery Other: No other concurrent anticancer agents No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2000-05; Primary Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fumoleau, MD, PhD, Study Chair — Centre Georges Francois Leclerc
Locations (11):
- U.Z. Gasthuisberg, Leuven, Belgium
- France (4):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lute Contre le Cancer,Georges-Francois Leclerc, Dijon
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Henri Becquerel, Rouen
- Rambam Medical Center, Haifa, Israel
- Azienda Ospedaliera di Padova, Padova (Padua), Italy
- Rotterdam Cancer Institute, Rotterdam, Netherlands
- Hospital Universitario 12 de Octubre, Madrid, Spain
- Switzerland (2):
  - Ospedale San Giovanni, Bellinzona
  - Clinique De Genolier, Genolier